CLINICAL TRIAL: NCT00826579
Title: Swiss Prospective, Multicenter Study Sentinel Lymph Node Procedure in Colon Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Rhein4031
Record Dates: First submitted 2009-01-13; First posted 2009-01-22 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2015-03

CONDITIONS: Colonic Neoplasms
Keywords: Sentinel lymph node; Lymph node analysis; Bone marrow analysis
MeSH Terms: conditions — Colonic Neoplasms | interventions — iso-sulfan blue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Colon cancer (Experimental): Colon cancer patients of all stages
  Interventions: Procedure: Sentinel lymph node procedure; Procedure: Bone marrow aspiration

INTERVENTIONS:
Procedure: Sentinel lymph node procedure — After careful mobilization of the affected colon segment, isosulfan blue 1% is injected in vivo into the subserosa circumferentially around the tumor. Lymph nodes in the mesentery staining blue within the first minutes are marked as SLN. The procedure is followed by a resection of the affected colon segment with standard lymphadenectomy.
  Other Names: Lymphazurin 1%, Ben Venue Labs Inc., Bedford OH
Procedure: Bone marrow aspiration — Prior to surgery, bone marrow is aspirated from both iliac crests. Bone marrow aspirates are analyzed for the presence of occult metastatic colon cancer cells.

SUMMARY:
The study is a feasibility and validation study of the sentinel lymph node (SLN) procedure in all stages of colon cancer. If the SLN can be reliably identified, it could be submitted to a more accurate histopathological examination (multiple sections, special staining). The detection of micrometastases in the SLN (occult stage III, upstaging) is possible. Patients with micrometastases should be considered at higher risk.

Additionally, a search for occult metastatic tumor cells in the bone marrow is performed.

ELIGIBILITY:
Inclusion Criteria:

* Colon cancer at any stage diagnosed histologically or high degree of suspicion for colon cancer at endoscopy, which cannot be confirmed with certainty in the biopsy. The diagnosis of cancer must be certain in the definitive histology.
* Possibility of transabdominal injection of the dye (cancers below the peritoneal reflection in which the injection of dye must be carried out through rectoscopy, are therefore excluded).
* Patient's informed consent

Exclusion Criteria:

* Prior intrabdominal tumor surgery
* Other preexisting malignancies
* Hypersensitivity/allergy to dye (isosulfan blue)
* Pregnancy
* Breast-feeding
* No patient's informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2000-05; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To assess the extent of upstaging due to the SLN procedure for colon cancer. | 1 month

SECONDARY OUTCOMES:
To evaluate the accuracy of the SLN procedure for colon cancer. To identify factors influencing the success of the procedure. To correlate SLN results with the presence of colon cancer cell in bone marrow aspirates. To assess OS and DFS. | 1 month, 3 and 5 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Carsten T. Viehl, MD, Principal Investigator — aktuell: Spitalzentrum Biel-Bienne; Markus Zuber, MD, Principal Investigator — Kantonsspital Olten
Locations (3):
- Switzerland (3):
  - Carsten T. Viehl, MD, Basel
  - Urban Laffer, MD, Biel
  - Markus Zuber, MD, Olten

REFERENCES:
- [Derived] Weixler B, Viehl CT, Warschkow R, Guller U, Ramser M, Sauter G, Zuber M. Comparative Analysis of Tumor Cell Dissemination to the Sentinel Lymph Nodes and to the Bone Marrow in Patients With Nonmetastasized Colon Cancer: A Prospective Multicenter Study. JAMA Surg. 2017 Oct 1;152(10):912-920. doi: 10.1001/jamasurg.2017.1514. PMID 28593306
- [Derived] Viehl CT, Guller U, Langer I, Laffer U, Oertli D, Zuber M. Factors influencing the success of in vivo sentinel lymph node procedure in colon cancer patients: Swiss prospective, multicenter study sentinel lymph node procedure in colon cancer. World J Surg. 2013 Apr;37(4):873-7. doi: 10.1007/s00268-013-1910-3. PMID 23354923